CLINICAL TRIAL: NCT04811677
Title: Comparison of a SegNet-based Algorithm Quantitatively Estimating Epifascial Fibrosis in Three-dimensional Computed Tomography Images to the Clinical Lymphedema Grading Method
Brief Title: Comparison of a SegNet-based Algorithm Estimating Epifascial Fibrosis
Status: Completed | Type: Observational
Sponsor: Chungnam National University Sejong Hospital (Other)
Responsible Party: Principal Investigator, Chang Ho Hwang, MD, PhD., Chief director, Chungnam National University Sejong Hospital
Other Study IDs: UUH 2018-04-009
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema | interventions — X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: radiology — image analysis

SUMMARY:
To approval for detecting lymphedema fibrosis before its progression, verification of CT-based quantification of suprafascial microscopic fibrosis has been tried.

DETAILED DESCRIPTION:
In lymphedema, proinflammatory cytokine-mediated progressive cascades always occur, leading to macroscopic fibrosis. However, no methods are practically available for measuring lymphedema-induced fibrosis before its deterioration. Technically, CT can visualize fibrosis in superficial and deep locations. For standardized measurement, verification of deep learning (DL)-based recognition was performed. A cross-sectional, observational cohort trial was conducted at a teaching university hospital. The protocol of this study was approved by the University Hospital Institutional Review Board and was registered at the Protocol Registration and Results System (PRS), www. clini caltr ials. gov (NCT04811677: https:// clini caltr ials. gov/ ct2/ show/ NCT04 811677? term= NCT04 81167 7& draw= 2& rank=1). All methods were performed in accordance with the relevant guidelines and regulations. The trial conformed to the tenets of the Declaration of Helsinki. Patients were included if they were clinically diagnosed with unilateral limb lymphedema and had undergone BEI analysis and CT scanning. The subjects provided written informed consent for publication of the case details. Data were collected as close to the CT scanning date as possible. Patients who were diagnosed with deep vein thrombosis, bilateral limb involvement, vascular disease, or local infection were excluded.

After narrowing window width of the absorptive values in CT images, SegNet-based semantic segmentation model of every pixel into 5 classes (air, skin, muscle/water, fat, and fibrosis) was trained (65%), validated (15%), and tested (20%). Then, 4 indices were formulated and compared with the standardized circumference difference ratio (SCDR) and bioelectrical impedance (BEI) results. In total, 2138 CT images of 27 chronic unilateral lymphedema patients were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* The patients who were clinically diagnosed with unilateral limb lymphedema and who underwent multi-frequency bio-electric impedance (BEI) analysis and CT scanning.

Exclusion Criteria:

* The patients who were diagnosed with deep vein thrombosis, bilateral limbs involvement, vascular diseases or local infection were excluded.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The patients who were clinically diagnosed with limb lymphedema.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
accuracy | within 1 week after CT scanning
  a ratio between the correctly classified pixel and all the classified pixel in one label.

SECONDARY OUTCOMES:
First index | within 1 week after CT scanning
  (P_(Fat in Affected)+P_(Fibrosis in Affected))/(P_(Fat in Unaffected)+P_(Fibrosis in Unaffected) ) " "

CONTACTS AND LOCATIONS:
Overall Officials: Chang Ho Hwang, Principal Investigator — Chungnam National University Sejong Hospital
Locations (1):
- Chungnam National University Sejong Hospital, Sejong, South Korea

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT04811677/SAP_000.pdf